CLINICAL TRIAL: NCT04216355
Title: The Feasibility of a Bridging Treatment With Low-dose Azacitidine (AZA) in Combination With Short Term CAG Derived Regimen Prior to Allogeneic Stem Cell Transplantation (Allo-HSCT) in Patients With Advanced Myelodysplastic Syndromes (MDS)
Brief Title: Low-dose AZA Combined With Short Term CAG Derived Regimen as a Bridging Treatment in Patients With Advanced MDS Prior to Allo-HSCT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Ting YANG, Principal Investigator, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDS-SCT-01
Record Dates: First submitted 2019-12-30; First posted 2020-01-02 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: MDS-EB
MeSH Terms: interventions — Azacitidine; CAG protocol

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AZA with CAG derived regimen (Experimental): Azacitidine 50mg/m²/day, D1-D5 (IV) Aclarubicin 5mg/m²/day, D1-D4 (IV) Cytarabine 10mg/m²/12h, D1-D6 (IV) G-CSF 5-10ug/kg/day, D1-D7 (SC)
  Interventions: Drug: Azacitidine; Drug: CAG Protocol

INTERVENTIONS:
Drug: Azacitidine — Low-dose AZA
Drug: CAG Protocol — Short term CAG derived regimen

SUMMARY:
This single arm, prospective study on the feasibility of a bridging treatment with low-dose azacitidine (AZA) in combination with short term CAG derived regimen prior to allogeneic stem cell transplantation (allo-HSCT) in patients with advanced myelodysplastic syndromes (MDS) .

ELIGIBILITY:
Inclusion Criteria:

* New Diagnosed advanced myelodysplastic syndrome (MDS) for whom an allogeneic hematopoietic stem cell transplant is planned
* Recipient of an allogeneic hematopoietic stem cell transplantation
* Age < 65 years
* ECOG performance status ≤2
* Written informed consent
* No psychological, familial, social, or geographic reason that would compromise clinical follow up

Exclusion Criteria:

* Relapsed or refractory advanced MDS
* Severe pshyciatric or organic disorder, supposed to be independent from advanced MDS, that would contraindicate treatment
* Known allergic or hypersensitivity to azacitidine, aclarubicin or cytarabine or to any of the test compounds, materials
* Concurrent, uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place the subject at unacceptable risk
* A co-morbid condition which, in the view of the Investigators, renders the subject at high risk from treatment complications

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Mean Time to Engraftment | Baseline to engraftment, assessed minimally 28 days post transplant

SECONDARY OUTCOMES:
Cumulative Incidence of Graft-versus Host Disease | Up to 2 years
Incidence of systemic infections | Up to 2 years
Overall survival | Up to 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China